CLINICAL TRIAL: NCT01911845
Title: An Open-label, Single-Arm, Phase 2 Study to Evaluate the Combination of ABT-450/r/ABT-267 and ABT-333 Coadministered With Ribavirin (RBV) in Adults With Genotype 1 Hepatitis C Virus (HCV) Infection Taking Methadone or Buprenorphine
Brief Title: An Open-label, Single Arm, Phase 2 Study to Evaluate ABT-450/r/ABT-267 and ABT-333 With Ribavirin (RBV) in Adults With Genotype 1 HCV Infection Taking Methadone or Buprenorphine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M14-103
Record Dates: First submitted 2013-05-13; First posted 2013-07-30 (Estimated); Results first posted 2015-01-06 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2015-08

CONDITIONS: Chronic Hepatitis C Infection; Chronic Hepatitis C
Keywords: HCV Genotype 1; Hepatitis Genotype 1; Interferon Free; methadone; HCV; Buprenorphine; Hepatitis C; Viekira Pak; paritaprevir; Viekira; ombitasvir; dasabuvir
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — paritaprevir; ombitasvir; dasabuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABT-450/r/ABT-267 and ABT-333, plus RBV (Experimental): ABT-450/r/ABT-267 (150/100/25 mg once daily) and ABT-333 (250 mg twice daily), plus weight-based ribavirin (RBV; 1,000 mg/day if <75 kg or 1,200 mg/day if ≥75 kg, divided twice daily) for 12 weeks
  Interventions: Drug: ABT-450/r/ABT-267; Drug: ABT-333; Drug: Ribavirin (RBV)

INTERVENTIONS:
Drug: ABT-450/r/ABT-267 — Tablet; ABT-450 coformulated with ritonavir and ABT-267
  Other Names: ABT-450 also known as paritaprevir; ABT-267 also known as ombitasvir
Drug: ABT-333 — Tablet
  Other Names: dasabuvir
Drug: Ribavirin (RBV) — Tablet

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of ABT-450/ritonavir/ABT-267 (ABT-450/r/ABT-267; ABT-450 also known as paritaprevir; ABT-267 also known as ombitasvir) and ABT-333 (also known as dasabuvir) coadministered with ribavirin (RBV) in hepatitis C virus (HCV) genotype 1-infected adults taking methadone or buprenorphine ± naloxone.

DETAILED DESCRIPTION:
This study consisted of 2 periods: a 12-week treatment period and a 48-week post-treatment period (for all participants who received study drugs). All participants who received at least 1 dose of study drug were to be followed for 48 weeks post-treatment to monitor for safety, HCV RNA, the emergence and/or persistence of resistant viral variants, and assessment of patient-reported outcome (PRO) instruments.

ELIGIBILITY:
Inclusion Criteria:

* Females must be practicing specific forms of birth control on study treatment, or be postmenopausal for more than 2 years or surgically sterile.
* Chronic HCV infection prior to study enrollment.
* Screening laboratory result indicating HCV genotype 1-infection.
* Subject must be treatment naive or previous pegylated interferon/ribavirin treatment experienced.
* Subjects must be on a stable opioid replacement therapy of methadone or buprenorphine ± naloxone for at least 6 months prior to screening.

Exclusion Criteria:

* Positive test result for Hepatitis B surface antigen (HBsAg) or anti-Human Immunodeficiency virus antibody (HIV Ab) at screening.
* Prior therapy with direct acting antiviral agents for the treatment of HCV, including telaprevir and boceprevir.
* Females who are pregnant or plan to become pregnant, or breastfeeding, or males whose partners are pregnant or planning to become pregnant within 7 months (or per local RBV label) after their last dose of study drug.
* Any current or past clinical evidence of cirrhosis such as ascites or esophageal varices, or prior biopsy showing cirrhosis, e.g., a Metavir Score of >3 or Ishak score of > 4.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Cohen, MD, Study Director — AbbVie

REFERENCES:
- [Result] Lalezari J, Sullivan JG, Varunok P, Galen E, Kowdley KV, Rustgi V, Aguilar H, Felizarta F, McGovern B, King M, Polepally AR, Cohen DE. Ombitasvir/paritaprevir/r and dasabuvir plus ribavirin in HCV genotype 1-infected patients on methadone or buprenorphine. J Hepatol. 2015 Aug;63(2):364-9. doi: 10.1016/j.jhep.2015.03.029. Epub 2015 Apr 1. PMID 25839406
- See also: Related Info — http://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ABT-450/r/ABT-267 and ABT-333, Plus RBV
Started | 38
Completed Study Drug | 37
Completed | 32
Not Completed | 6
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 1
Not completed — Other (not specified) | 3

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Arm/Group | ABT-450/r/ABT-267 and ABT-333, Plus RBV
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment
Description: The percentage of participants with sustained virologic response (plasma hepatitis C virus ribonucleic acid [HCV RNA] level less than the lower limit of quantification [< LLOQ]) 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after the last actual dose of study drug
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ABT-450/r/ABT-267 and ABT-333, Plus RBV
Number analyzed (Participants) | 38
Percentage of participants | 97.4 [92.3 to 100]

2. Secondary Outcome: Percentage of Participants With Virologic Failure During Treatment
Description: Virologic failure during treatment was defined as rebound (confirmed HCV RNA greater than or equal to the lower limit of quantitation [≥ LLOQ] after HCV RNA < LLOQ during treatment, or confirmed increase from the lowest value post baseline in HCV RNA [2 consecutive HCV RNA measurements > 1 log(subscript)10(subscript) IU/mL above the lowest value post baseline] at any time point during treatment) or fail to suppress (HCV RNA ≥ LLOQ) persistently during treatment with at least 6 weeks [≥ 36 days] of treatment.
Time Frame: Baseline (Day 1), and Treatment Weeks 1, 2, 4, 6, 8, 10, and 12
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | ABT-450/r/ABT-267 and ABT-333, Plus RBV
Number analyzed (Participants) | 38
Percentage of participants | 0

3. Secondary Outcome: Percentage of Participants With Virologic Relapse Post-treatment
Description: Participants were considered to have virologic relapse after treatment if they had confirmed quantifiable plasma Hepatitis C virus ribonucleic acid (HCV RNA) ≥ lower limit of quantification (LLOQ) between the end of treatment and 12 weeks after the last dose of study drug among participants who completed treatment with HCV RNA < LLOQ at the end of treatment. Completion of treatment was defined as a study drug duration ≥ 77 days.
Time Frame: From the end of treatment through 12 weeks after the last actual dose of study drug
Population: All randomized participants who received at least 1 dose of study drug with HCV RNA < LLOQ at the final treatment visit who completed treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | ABT-450/r/ABT-267 and ABT-333, Plus RBV
Number analyzed (Participants) | 37
Percentage of participants | 0

4. Secondary Outcome: Area Under the Plasma Concentration-time Curve (AUC) for ABT-450, Ritonavir, ABT-267, ABT-333, ABT-333 M1 Metabolite, and Ribavirin
Description: Blood samples were collected pre-dose (time 0) and at 2, 4, 6, and 24 hours post-dose at one visit between treatment week 2 and treatment week 12, and were analyzed using validated analytical methods. A total of 22/38 participants consented for intensive pharmacokinetic blood sampling. Area under the plasma concentration-time curve from time 0 to 24 hours (AUC24 in ng*hr/mL)] was estimated using noncompartmental analyses. For ABT-450, ritonavir, and ABT-267, the AUC from time 0 to the last measureable concentration (AUCt in ng*hr/mL) was calculated instead of AUC24 due to time deviations at 24 hours. The AUCt values are approximately equivalent to AUC24. For ABT-333, ABT-333 M1, and RBV, the AUC from time 0 to 12 hours (AUC12 in ng*hr/mL) after the morning dose was calculated using the 24-hour concentration as the 12-hour concentration as dosing was twice a day and a 12-hour sample was not collected in this study.
Time Frame: Pre-dose (time 0) and 2, 4, 6, and 24 hours post-dose
Population: Participants who consented for intensive pharmacokinetic blood sampling
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Buprenorphine ± Naloxone: Participants were on a stable opioid replacement therapy of buprenorphine ± naloxone during the Treatment Period, and for at least six months prior to screening.
- Methadone: Participants were on a stable opioid replacement therapy of methadone during the Treatment Period, and for at least six months prior to screening.
Arm/Group | Buprenorphine ± Naloxone | Methadone
Number analyzed (Participants) | 12 | 10
ng*hr/mL
  ABT-450 | 27438.94 (34380.77) | 37174.89 (49655.37)
  Ritonavir | 14303.27 (8367.86) | 11375.38 (5586.62)
  ABT-267 | 1523.48 (4444.58) | 1486.72 (519.84)
  ABT-333 | 5666.15 (2550.86) | 5021.41 (2353.06)
  ABT-333 M1 metabolite | 3086.73 (1807.51) | 2950.36 (2094.61)
  Ribavirin | 33362.24 (10340.16) | 33499.39 (10697.75)

5. Secondary Outcome: Maximum Plasma Concentration (Cmax) for ABT-450, Ritonavir, ABT-267, ABT-333, ABT-333 M1 Metabolite, and Ribavirin
Description: Blood samples were collected pre-dose (time 0) and at 2, 4, 6, and 24 hours post-dose at one visit between treatment week 2 and treatment week 12, and were analyzed using validated analytical methods. A total of 22/38 participants consented for intensive pharmacokinetic blood sampling. Maximum plasma concentration (Cmax; measured in ng/mL) was directly determined from the concentration-time data.
Time Frame: Pre-dose (time 0) and 2, 4, 6, and 24 hours post-dose
Population: Participants who consented for intensive pharmacokinetic blood sampling
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Buprenorphine ± Naloxone | Methadone
Number analyzed (Participants) | 12 | 10
ng/mL
  ABT-450 | 3269.50 (4388.48) | 2973.30 (3371.83)
  Ritonavir | 1261.92 (657.35) | 888.70 (409.56)
  ABT-267 | 102.00 (27.21) | 95.98 (35.56)
  ABT-333 | 805.08 (354.04) | 671.90 (302.08)
  ABT-333 M1 metabolite | 469.92 (271.13) | 439.64 (272.91)
  Ribavirin | 3389.17 (1064.98) | 3232.00 (948.39)

6. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) for ABT-450, Ritonavir, ABT-267, ABT-333, ABT-333 M1 Metabolite, and Ribavirin
Description: Blood samples were collected pre-dose (time 0) and at 2, 4, 6, and 24 hours post-dose at one visit between treatment week 2 and treatment week 12, and analyzed using validated analytical methods. A total of 22/38 participants consented for intensive pharmacokinetic blood sampling. The time to maximum plasma concentration (Tmax; measured in hours) was directly determined from the concentration-time data.
Time Frame: Pre-dose (time 0) and 2, 4, 6, and 24 hours post-dose
Population: Participants who consented for intensive pharmacokinetic blood sampling
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Buprenorphine ± Naloxone | Methadone
Number analyzed (Participants) | 12 | 10
hours
  ABT-450 | 4.38 (1.45) | 6.81 (6.04)
  Ritonavir | 4.18 (1.33) | 7.01 (5.97)
  ABT-267 | 4.69 (1.00) | 5.26 (0.98)
  ABT-333 | 4.25 (2.74) | 4.05 (1.40)
  ABT-333 M1 metabolite | 4.40 (0.84) | 4.65 (1.11)
  Ribavirin | 3.72 (2.95) | 5.83 (4.34)

7. Secondary Outcome: Plasma Trough Concentration (Ctrough) for ABT-450, Ritonavir, ABT-267, ABT-333, ABT-333 M1 Metabolite, and Ribavirin
Description: Blood samples were collected pre-dose (time 0) and at 2, 4, 6, and 24 hours post-dose at one visit between treatment week 2 and treatment week 12, and analyzed using validated analytical methods. A total of 22/38 participants consented for intensive pharmacokinetic blood sampling. Minimum plasma concentration (C trough; measured in ng/mL) was directly determined from the concentration-time data.
Time Frame: Pre-dose (time 0) and 2, 4, 6, and 24 hours post-dose
Population: Participants who consented for intensive pharmacokinetic blood sampling
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Buprenorphine ± Naloxone | Methadone
Number analyzed (Participants) | 12 | 10
ng/mL
  ABT-450 | 170.01 (368.36) | 458.53 (988.11)
  Ritonavir | 167.35 (406.50) | 136.87 (273.44)
  ABT-267 | 33.75 (17.28) | 32.78 (14.11)
  ABT-333 | 223.76 (246.63) | 147.95 (115.20)
  ABT-333 M1 metabolite | 86.98 (110.35) | 71.10 (83.23)
  Ribavirin | 2555.83 (1115.82) | 2632.00 (1039.54)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of study drug administration until 30 days after the last dose, up to 16 weeks. Serious adverse events were collected from the time of informed consent until the end of participation in the study (65 weeks).
Arm/Group | ABT-450/r/ABT-267 and ABT-333, Plus RBV
Serious Adverse Events (participants affected / at risk) | 2/38
Other Adverse Events (participants affected / at risk) | 35/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-450/r/ABT-267 and ABT-333, Plus RBV (N=38)
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-450/r/ABT-267 and ABT-333, Plus RBV (N=38)
ANAEMIA (Blood and lymphatic system disorders) | 4
ABDOMINAL PAIN (Gastrointestinal disorders) | 2
DIARRHOEA (Gastrointestinal disorders) | 3
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 3
GINGIVAL PAIN (Gastrointestinal disorders) | 2
NAUSEA (Gastrointestinal disorders) | 19
VOMITING (Gastrointestinal disorders) | 4
FATIGUE (General disorders) | 18
IRRITABILITY (General disorders) | 4
OEDEMA PERIPHERAL (General disorders) | 2
PYREXIA (General disorders) | 3
NASOPHARYNGITIS (Infections and infestations) | 3
ORAL HERPES (Infections and infestations) | 2
TOOTH ABSCESS (Infections and infestations) | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2
HAEMOGLOBIN DECREASED (Investigations) | 2
DECREASED APPETITE (Metabolism and nutrition disorders) | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 3
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2
DIZZINESS (Nervous system disorders) | 2
HEADACHE (Nervous system disorders) | 12
MIGRAINE (Nervous system disorders) | 2
PARAESTHESIA (Nervous system disorders) | 2
ANXIETY (Psychiatric disorders) | 5
CONFUSIONAL STATE (Psychiatric disorders) | 2
DEPRESSION (Psychiatric disorders) | 3
INSOMNIA (Psychiatric disorders) | 7
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2
RASH (Skin and subcutaneous tissue disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.